CLINICAL TRIAL: NCT05673720
Title: Feasibility, Acceptability, and Preliminary Efficacy of Combined Transcranial Direct Current Stimulation and Mindfulness for Pain After Total Knee Arthroplasty
Brief Title: Brain Stimulation and Meditation for Pain After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Geraldine Martorella, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00003476; 140009-140 (Other Grant/Funding Number: Florida State University)
Record Dates: First submitted 2022-12-19; First posted 2023-01-06 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- preoperative active tDCS+MBI (Experimental): Active tDCS with simultaneous meditation intervention will be applied.
  Interventions: Device: active tDCS paired with active MBM
- preoperative sham tDCS+MBI (Sham Comparator): Sham tDCS with simultaneous sham MBM intervention will be delivered.
  Interventions: Device: sham tDCS paired with sham MBM

INTERVENTIONS:
Device: active tDCS paired with active MBM — Active tDCS with a constant current intensity of 2 milli ampere( mA)will be applied for 20 minutes per session for 5 times via the Soterix 1x1 tDCS mini-CT Stimulator device with headgear and saline-soaked surface sponge electrodes. The meditation intervention will be applied simultaneously with tDCS for 20 minutes per session for 5 times by a recorded meditation.
  Arms: preoperative active tDCS+MBI
Device: sham tDCS paired with sham MBM — For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds. The sham MBM intervention will be delivered via a CD player that will look identical in both active and sham MBM.
  Arms: preoperative sham tDCS+MBI

SUMMARY:
Feasibility, acceptability, and preliminary efficacy of combined transcranial direct current stimulation and mindfulness for pain after total knee arthroplasty

DETAILED DESCRIPTION:
The project is to assess the preliminary feasibility, acceptability, and efficacy of self-administered preoperative tDCS+MBI in older adults (50+) undergoing TKR. And to determine the effects of 5, 20-minute preoperative self-administered tDCS sessions combined with brief MBI on analgesic medication consumption following TKR.

ELIGIBILITY:
Inclusion Criteria:

* elective unilateral knee total replacement
* mentally capable of reading, giving consent and following instructions
* being able to answer questions in English
* not pregnant

Exclusion Criteria:

* history of brain surgery, brain tumor, seizure, stroke, or intracranial metal implantation
* systemic rheumatic disorders, including rheumatoid arthritis, systemic lupus erythematosus, and fibromyalgia
* alcohol/substance abuse
* current use of sodium channel blockers, calcium channel blockers and NMDS receptor antagonists
* hospitalization within the preceding year for psychiatric illness
* no access to a device with internet access that can be used for secure videoconferencing for real-time remote supervision

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic, Tallahassee, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 2023 and February 2024. Participants were recruited at their preoperative visit. A clinician or a research coordinator from the clinic conducted a pre-screening of potentially eligible participants, and introduced the study to potential participants at their preoperative visit. If the individual agreed to learn more, the PI or RA entered the room to discuss study, answer questions and scheduled an appointment.
Pre-assignment Details: A total of 40 potential participants were approached. Of these, 8 (20%) did not meet inclusion criteria (e.g., partial replacement surgery, fibromyalgia) and 8 declined to participated (20%) mainly because they were living too far to travel to the lab for the baseline and last appointments before surgery.
Groups:
- Preoperative Active tDCS+MBI: Active tDCS with simultaneous meditation intervention will be applied for 20 minutes X 5 sessions.
- Preoperative Sham tDCS+MBI: Sham tDCS with simultaneous sham MBM intervention will be delivered for 20 minutes X 5 sessions.
Period: Overall Study
Arm/Group | Preoperative Active tDCS+MBI | Preoperative Sham tDCS+MBI
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative Active tDCS+MBI | Preoperative Sham tDCS+MBI | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — age
  years | 67.4 (9.7) | 67.1 (9.3) | 67.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: Participants]
  United States | 12 | 12 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 3 | 1 | 4
  White | 8 | 11 | 19
  multiple ethnicity | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Consumption
Description: The dose of every opioid received within 3 days postoperatively will be transcribed and converted into standardized parenteral morphine equivalents using the Centers for Disease and Control Prevention Guidelines on opioids. A total in milligrams will be calculated for each day and means will be obtained for all groups.
Time Frame: day 3 after surgery
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Preoperative Active tDCS+MBI | Preoperative Sham tDCS+MBI
Number analyzed (Participants) | 12 | 12
mg | 0 (0) | 0 (0)

2. Secondary Outcome: Numerical Rating Scale (NRS)
Description: The NRS total score ranges from 0 (no pain) to 10 (most intense pain imaginable).
Time Frame: day 3 after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preoperative Active tDCS+MBI | Preoperative Sham tDCS+MBI
Number analyzed (Participants) | 12 | 12
units on a scale | 6.18 (1.40) | 5.71 (2.56)

3. Secondary Outcome: Brief Pain Inventory (BPI)
Description: It includes seven items and evaluates the impact of pain on general activity, mood, walking, work, relationships, sleep, and enjoyment of life via a NRS (0-10). Each item represents a subscale and can be scored and analyzed individually (0-10), with the anchors being "does not interfere" (0) and "completely interferes" (10). A total interference score can also be calculated by taking the sum of all the items (score range 0-70). A higher score reflects worse outcomes : higher pain interference with activities.
Time Frame: day 3 after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preoperative Active tDCS+MBI | Preoperative Sham tDCS+MBI
Number analyzed (Participants) | 12 | 12
units on a scale | 6.04 (2.17) | 5.51 (3.39)

4. Secondary Outcome: Patient Health Questionnaire-4 (PHQ-4)
Description: The PHQ-4 has a total score range of 0-12, which is broken down into four ranges: normal (0-2), mild (3-5), moderate (6-8), and severe (9-12) psychological distress. For the subscales (PHQ-2 for depression and GAD-2 for anxiety), the score range is 0-6. higher values represent a worse outcome
Time Frame: day 3 after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preoperative Active tDCS+MBI | Preoperative Sham tDCS+MBI
Number analyzed (Participants) | 12 | 12
units on a scale | 5.4 (2.76) | 8.0 (3.6)

5. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: to assess patients' pain-related catastrophic thoughts. It includes 13 items divided into three subscales: rumination (4 items), magnification (3 items), and helplessness (6 items). Each item is rated on a 5-point scale with the end points not at all (score=0) and all the time (score=4). The total score range for the Pain Catastrophizing Scale (PCS) is 0 to 52, where a higher score indicates greater levels of pain catastrophizing.
Time Frame: day 3 after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preoperative Active tDCS+MBI | Preoperative Sham tDCS+MBI
Number analyzed (Participants) | 12 | 12
units on a scale | 20.56 (7.76) | 25.25 (13.05)

ADVERSE EVENTS:
Time Frame: from baseline up to one month
Description: questionnaire after each session + self-report to research assistant during study regarding serious and adverse events
Arm/Group | Preoperative Active tDCS+MBI | Preoperative Sham tDCS+MBI
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoperative Active tDCS+MBI (N=12) | Preoperative Sham tDCS+MBI (N=12)
tingling (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)

LIMITATIONS AND CAVEATS:
we had fNIRS malfunction at the beginning of the study and did not include cortical activity as an outcome in this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT05673720/Prot_001.pdf
  • Statistical Analysis Plan (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT05673720/SAP_004.pdf
  • Informed Consent Form (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT05673720/ICF_000.pdf